CLINICAL TRIAL: NCT00108511
Title: Effect of Gemfibrozil on Serum GPI Phospholipase D and Triglycerides
Brief Title: Effect of Gemfibrozil on Serum Glycosylphosphatidylinositol (GPI) Phospholipase D and Triglycerides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CLNB-009-04S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; lipoproteins; triglycerides; serum GPI-PLD (glycosylphosphatidylinositol-specific phospholipase D)
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Gemfibrozil

INTERVENTIONS:
Drug: Gemfibrozil

SUMMARY:
The purpose of this study is to examine the role of glycosylphosphatidylinositol-specific phospholipase D (GPI-PLD) in triglyceride metabolism.

DETAILED DESCRIPTION:
Increased fasting serum triglyceride levels are associated with an increased risk of coronary artery disease. However, triglyceride levels in the postprandial state are a more sensitive marker of coronary artery disease. Postprandial elevations in triglycerides result from a decrease in the catabolism of triglyceride-rich lipoproteins, i.e. chylomicrons and very low density lipoproteins (VLDL). This leads to an accumulation of atherogenic remnants of triglyceride-rich lipoproteins. Although fasting triglycerides are the best predictors of postprandial triglycerides, differences in fasting triglycerides only partially account for the variation in magnitude of postprandial triglycerides. Recently, we have identified a new protein involved in triglyceride-rich lipoprotein catabolism, glycosylphosphatidylinositol-specific phospholipase D (GPI-PLD). We have shown that elevated levels of GPI-PLD are associated with increased fasting triglyceride levels. Serum GPI-PLD is associated with high density lipoproteins (HDL) in the fasting state and exchange onto VLDL in the postprandial state. Hepatic GPI-PLD decreases triglyceride-rich lipoprotein catabolism in the liver. Hepatic and serum GPI-PLD levels are decreased by peroxisome proliferator receptor (PPAR) alpha agonist treatment, which also reduces fasting and postprandial triglycerides. The central hypothesis of this application is that variations in GPI-PLD expression account for a portion of the differences in fasting and postprandial triglycerides among humans.

The objective of this proposal is to determine the role of GPI-PLD in regulating fasting triglycerides and post-prandial hypertriglyceridemia in humans. This will be accomplished by conducting a double blind, placebo controlled study in humans examining the effect of gemfibrozil on fasting and postprandial triglycerides in relationship to the variation and changes in GPI-PLD before and after gemfibrozil.

Our specific objectives are:

* 1a) Determine the extent to which variations in GPI-PLD account for differences in fasting and postprandial triglycerides
* 1b) Establish the degree to which the lowering of fasting and postprandial triglycerides by gemfibrozil is accounted for by changes in GPI-PLD.
* 2) Quantify the changes in serum GPI-PLD and distribution of GPI-PLD among lipoproteins in the postprandial state.

This will be the first prospective bench-to-bedside study examining the role of GPI-PLD in triglyceride metabolism. This proposal will be the first in humans examining 1) the role of a novel protein, GPI-PLD, in triglyceride metabolism, and 2) the effect of gemfibrozil, a drug currently used clinically to lower triglyceride levels, on GPI-PLD levels in humans. It is expected that the results from this study will increase our understanding of triglyceride metabolism and develop new information in understanding the regulation of GPI-PLD and its relationship to triglyceride metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <75
* Fasting triglycerides >150 mg/dl

Exclusion Criteria:

* Fasting triglycerides >600 mg/dl
* LDL >130 mg/dl
* Concurrent lipid lowering therapy
* Known hypersensitivity to gemfibrozil
* Alcohol intake >30 gm/day (2 drinks/day)
* Fasting glucose >125 mg/dl or known type 2 diabetes
* AST or ALT > 2.0 x upper limit of normal
* Creatinine: men >1.4 mg/dl, women >1.3 mg/dl
* Cancer treatment in the past 5 years (unless cured)
* Infectious diseases including HIV or tuberculosis
* Significant cardiac disease in the past 6 months (myocardial infarction, coronary artery bypass graph, angioplasty, class 3 or 4 congestive heart failure, left bundle branch block, third degree AV block)
* Uncontrolled hypertension (systolic blood pressure [SBP] >180 or diastolic blood pressure [DBP] > 105 mm Hg)
* Anemia (hematocrit <40% men, <35% women)
* Any other significant systemic disease or medication that could interfere with tolerance of medication or outcome
* Any indication that a participant will be unable to adhere to the protocol
* Unable to give informed consent
* Pregnant or breastfeeding females or a female who plans to become pregnant while participating in the study

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Locations (1):
- Roudebush VA Medical Center, Indianapolis, Indiana, United States